CLINICAL TRIAL: NCT06950879
Title: Implicit Central Hand Representation in Children With Neonatal Brachial Plexus Palsy: Interrater and Intrarater Reliability of the HandUZ Device - A Validation Study
Brief Title: Validation Study Of A Digital Measuring Device For Central Hand Representation In Children With A Neonatal Brachial Plexus Palsy
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0515
Record Dates: First submitted 2025-04-18; First posted 2025-04-30 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Brachial Plexus Palsy
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: A group of 20 children aged 8-18 with a neonatal brachial plexus palsy. We measured the implicit map of hand size 6 times for each hand.
  Interventions: Other: Measurement

INTERVENTIONS:
Other: Measurement — A wooden construction was built consisting of two plates with dimensions of 35 x 29 cm: a bottom plate, with a measuring mat glued to it, a movable middle plate and a smaller top plate, allowing to mount a standardized overhead camera.
  Participants were seated and placed one hand palm down on the measuring mat on the bottom plate. The hand was aligned with the midline of the body, lay flat with the fingers straight and lightly spread. First the actual landmarks were marked on the computer. Subsequently the participants hand was occluded by adding the middle plate. Participants were verbally cued to mark a certain landmark with their contralateral hand. These indicated points were marked on the computer. Before and after each trial, a picture was taken without the occluding board to ensure that the hand had not moved from its original position by digitally overlaying the images

SUMMARY:
Hand function is one of the most complex and sophisticated sensorimotor skills, controlled by the interplay of precise motor efferent and multisensory afferent stimuli. A coherent central representation of the hand is essential for performing hand movements in a changing environment.

However, the hand representation in the brain consists of many modalities (visual, proprioceptive, anthropometric,...). The division between explicit (conscious) and implicit (unconscious) representation of the hand is accepted by a large group of researchers. The explicit representation of the hand is based partly on visual afferents, the implicit on all other afferent inputs.

Impaired hand function in everyday use after injury may be due to aberrant hand representation. Previous research showed that children with neonatal brachial plexus injury have impaired implicit hand representation with respect to hand size. Despite the good reproducibility of test results reported in the literature, the measurement method is very cumbersome.

In the current technological revolution, digitalisation of the device is the ideal solution to make the measurement method clinically applicable in daily practice.

Therefore, a new prototype digital device has been developed to automate the measurement method. This prototype works on the same principle and has the same dimensions as previous studies. It includes digital storage and processing of the measurement results. This study investigates the reproducibility (inter- and intra-observer) of the digital prototype.

The study will recruit children aged between 8 and 18 years with a neonatal brachial plexus injury.

Doctors treating this patient group will explain the study during consultations and provide a flyer. Participation in the study means that the patient will be invited to the UZ Ghent Paediatric Rehabilitation Centre, where two different doctors will independently perform the measurement. Specifically, they will be asked to place their hand on a mat and the fingertips, knuckles and wrist will be marked on the device. A wooden board is then placed over the hand so that the hand is no longer visible. The subject is then asked to indicate the fingertips, knuckles and wrist in random order, again recorded on the device. The test takes 5 to a maximum of 10 minutes (depending on cooperation). This measurement is repeated a 6 times on each hand.

Based on these measurements, the device calculates the average of each participant's perceived hand width and finger length. These values are compared with the actual hand width and finger length. This allows us to calculate a percentage of overestimation. Studies using such data have already been published.

The aim of this study is to measure the reproducibility (inter- and intraobserver) of the digitised version.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a Neonatal Brachial Plexus Palsy

Exclusion Criteria:

* Presence of any other important locomotor, neurological or psychiatric disorder

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between the age of 8 and 18 with a Neonatal Brachial Plexus Palsy
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van der Looven R, Hermans L, Coupe AM, De Muynck M, Vingerhoets G. Neonatal brachial plexus palsy and hand representation in children and young adults. Dev Med Child Neurol. 2022 Feb;64(2):183-191. doi: 10.1111/dmcn.15008. Epub 2021 Aug 17. PMID 34405401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between Januari and April 2025 at the Child Rehabilitation Centre of Ghent University Hospital. Eligible children with a confirmed diagnosis of neonatal brachial plexus palsy (NBPP) were identified during regular consultations at the multidisciplinary NBPP clinic. Information about the study was provided verbally and in writing to families. A total of 18 participants aged 8- 18 were included.
Groups:
- Participants: A group of 18 children aged 8-18 with a neonatal brachial plexus palsy.
Period: Overall Study
Arm/Group | Participants
Started | 18 (Each participant underwent six trials per hand using the HandUZ device. Implicit finger length was estimated for both left and right hands, resulting in multiple measurement units per participant. However, only full participants were considered as the unit of assignment and analysis in this study. One participant could not complete any measurement due to motor limitations and was excluded from analysis.)
Completed | 17
Not Completed | 1
Not completed — Unable to complete task due to motor impairment | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants: 17 children aged 8-18 with a neonatal brachial plexus palsy.
Arm/Group | Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Intrarater Reliability of Implicit Finger Length Estimates Using the HandUZ Device
Description: Intrarater reliability was assessed using the intraclass correlation coefficient (ICC[3,1]) based on two sets of averaged finger length estimates (FL) per participant, measured across two time points by the same rater. FL was calculated in centimeters as the Euclidean distance between the fingertip and metacarpophalangeal (MCP) joint for each digit. Data were averaged across fingers and hands to yield a single participant-level value. ICCs were calculated using a two-way mixed-effects model, absolute agreement. A higher ICC indicates greater measurement reliability. Each participant contributed two independent values (left and right hand), but the unit of analysis is the participant. Results for both hands are reported in separate rows.
Time Frame: Single session (approximately 45 minutes)
Measure: Number (95% Confidence Interval); unit: Intraclass Correlation Coefficient
Groups:
- Participants: A group of 17 children aged 8-18 with a neonatal brachial plexus palsy. We measured the implicit map of hand size 6 times for each hand.
Arm/Group | Participants
Number analyzed (Participants) | 17
Intraclass Correlation Coefficient
  Left hand | 0.91 [0.75 to 0.96]
  Right hand | 0.92 [0.67 to 0.98]

2. Secondary Outcome: Interrater Reliability of Implicit Finger Length Estimates Using the HandUZ Device
Description: Interrater reliability was assessed using the intraclass correlation coefficient (ICC[3,1]) based on two sets of averaged finger length estimates (FL) measured independently by two trained raters. FL was computed per finger (in cm) as the Euclidean distance between fingertip and MCP joint using HandUZ software. Values were averaged across fingers and hands. ICCs were calculated using a two-way mixed-effects model, absolute agreement. Separate ICC values are provided for the left and right hands in the results table, but both are reported under this single outcome measure. Each participant contributed two independent values (left and right hand), but the unit of analysis is the participant. Results for both hands are reported in separate rows
Time Frame: Single session (approximately 45 minutes)
Measure: Number (95% Confidence Interval); unit: Intraclass Correlation Coefficient
Arm/Group | Participants
Number analyzed (Participants) | 17
Intraclass Correlation Coefficient
  Left hand | 0.72 [0.27 to 0.90]
  Right hand | 0.71 [0.36 to 0.88]

ADVERSE EVENTS:
Time Frame: During single testing session (approximately 45 minutes)
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT06950879/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT06950879/SAP_001.pdf
  • Informed Consent Form (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT06950879/ICF_002.pdf